CLINICAL TRIAL: NCT01074424
Title: Development of a Serum Proteomic Profile for Cervical Cancer With Potential Prognostic Value
Brief Title: Studying Biomarkers in Blood Samples From Patients With Invasive Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Philip J. DiSaia, Gynecologic Oncology Group
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000665346; GOG-8006
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Cervical Cancer
Keywords: stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

INTERVENTIONS:
Genetic: proteomic profiling
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is looking at biomarkers in blood samples from patients with invasive cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To develop a serum proteomic profile for cervical cancer using banked pre-treatment serum specimens from patients with invasive cervical cancer and to determine if this serum proteomic profile has possible utility in cervical cancer prognosis.

Secondary

* To develop a serum proteomic profile for cervical cancer using banked post-treatment serum specimens from these patients and to determine if this serum proteomic profile has possible utility in cervical cancer prognosis.

OUTLINE: This is a multicenter study.

Banked serum specimens are used to generate proteomic profiles.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma, squamous cell carcinoma, or adenosquamous cell carcinoma of the cervix

  * Stage IIB, III, or IVA disease
* Eligible and evaluable for GOG-0191
* Pre- and/or post-treatment serum specimens available for proteomic analysis

PATIENT CHARACTERISTICS:

* Patient has given consent to allow their specimen(s) to be used for future cancer research

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Generation of a serum proteomic profile using banked pre-treatment serum specimens that may have potential utility for cervical cancer prognosis (overall survival and progression-free survival [PFS])

SECONDARY OUTCOMES:
Generation of a serum proteomic profile using banked post-treatment serum specimens that may have potential utility for cervical cancer prognosis (overall survival and PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Samir N. Khleif, MD, Principal Investigator — National Cancer Institute (NCI)